CLINICAL TRIAL: NCT00100139
Title: A Randomized Two-Period Crossover, Clinical Bioequivalence Study Comparing the Pharmacokinetics of Liposome Entrapped Paclitaxel Easy to Use (LEP-ETU) Formulation Versus Taxol® in Patients With Advanced Cancer
Brief Title: Comparison of Liposome Entrapped Paclitaxel Easy to Use (LEP-ETU) and Taxol® Pharmacokinetics in Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: INSYS Therapeutics Inc (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LEP-ETU-102A
Record Dates: First submitted 2004-12-23; First posted 2004-12-24 (Estimated); Last update posted 2011-07-04 (Estimated); Status verified 2011-06

CONDITIONS: Neoplasm
Keywords: Neoplasm; Cancer; NeoPharm; Liposomes; Taxol; Paclitaxel; Anti-cancer; Advanced neoplasm; Advanced cancer; Chemotherapy; Refractory cancer; Metastatic cancer
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — Paclitaxel; Injections

INTERVENTIONS:
Drug: Liposome Entrapped Paclitaxel Easy to Use (LEP-ETU)
Drug: Paclitaxel for injection (Taxol)

SUMMARY:
In this study, Liposome Entrapped Paclitaxel Easy to Use (LEP-ETU) is being compared to Taxol® to examine whether the paclitaxel in these 2 formulations undergoes similar processing by the body. Safety and tolerability of LEP-ETU and Taxol will also be assessed. In this study, each patient will receive one intravenous infusion of LEP-ETU or Taxol, followed 3 weeks later by an infusion of the other drug, at the same dose and infusion duration. Multiple blood samples will be taken for analysis before, during, and after both drug infusions. Upon completing these 2 Cycles of treatment, eligible patients may enroll in an extension study (LEP-ETU-102B) to continue treatment with LEP-ETU.

LEP-ETU is a liposomal formulation of paclitaxel, a widely used anti-cancer drug. This LEP-ETU formulation of paclitaxel is being developed to potentially reduce toxicities associated with Taxol, by eliminating the drug formulation component polyoxyethylated castor oil (Cremophor® EL). In LEP-ETU, paclitaxel is associated with liposomes, which are microscopic membrane-like structures created from lipids (fats). Thus, the LEP-ETU formulation could potentially have reduced toxicity, while maintaining or enhancing efficacy.

DETAILED DESCRIPTION:
This Phase 1B, open-label, two-period crossover bioequivalence study is designed to compare the pharmacokinetics (PK) of LEP-ETU and Taxol in patients with advanced cancer. Patients are randomized to determine which drug is administered first. A single dose of LEP-ETU or Taxol (Cycle A) will be administered, followed 3 weeks later by a single dose of the other drug (Cycle B). Blood samples for PK analysis will be taken before, during, and after the infusion of each drug. Following successful completion of both Cycles in this study, patients may be eligible for additional cycles of treatment with LEP-ETU in the LEP-ETU-102B extension study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have advanced histologically diagnosed non-hematological malignancy for which there is no curative therapy and for which treatment with single agent paclitaxel is appropriate in the opinion of the investigator.
* Patients must have a life expectancy of 12 weeks or more.
* Patients must have an ECOG Performance Status of 0-2.
* Patients must have recovered from acute toxicities of prior treatment. Specifically: *4 or more weeks must have elapsed since receiving any investigational agent. *3 or more weeks must have elapsed since receiving any radiotherapy, or treatment with cytotoxic or biologic agents (6 weeks or more for mitomycin or nitrosureas). Chronic treatment with non-investigational gonadotropin-releasing hormone analogs or other hormonal or supportive care is permitted. *2 or more weeks must have elapsed since any prior surgery or granulocyte-stimulating growth factor therapy.

  * Patients must be in adequate condition as evidenced by the following clinical laboratory values: *Absolute neutrophil count (ANC) ≥1,500/mm³, *Platelet count ≥100,000/mm³, *Hemoglobin ≥9.0 g/dL, *Albumin ≥3.0 g/dl, *Serum creatinine ≥2.0 mg/dL, *Total bilirubin 1.5 x the institutional upper limit of normal (ULN) or greater. *Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 x ULN. In the case of known liver metastasis, ALT and AST ≤5 x ULN. *Alkaline phosphatase (ALP) ≤2.5 x ULN. No ULN applies to alkaline phosphatase in the case of known bone metastasis.
  * Patients (male and female) must be willing to practice an effective method of birth control during the study.
  * Patients must be available for and able to comply with the study-specific blood sampling requirements for pharmacokinetic evaluations.
  * Patients or legal representative must understand the investigational nature of this study and sign an Institutional Review Board (IRB) approved written informed consent form prior to treatment.

Exclusion Criteria:

* Active uncontrolled bleeding or bleeding diathesis (e.g., active peptic ulcer disease).
* Any active infection requiring parenteral or oral antibiotic treatment; any use of trimethoprim, including use for antimicrobial prophylaxis.
* Known infection with human immunodeficiency virus (HIV) or hepatitis virus.
* Active heart disease including myocardial infarction or congestive heart failure within the previous 6 months, symptomatic coronary artery disease, or arrhythmias currently requiring medication.
* Known or suspected active central nervous system metastasis. (Patients stable 8 weeks after completion of treatment for central nervous system metastasis are eligible.)
* Impending or symptomatic spinal cord compression or carcinomatous meningitis.
* Having pre-existing clinically significant neuropathy (National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) greater than or equal to Grade 2 neuromotor or Grade 2 neurosensory) except for abnormalities due to cancer.
* Having known hypersensitivity to paclitaxel or liposomes.
* Receiving any agent that could interfere with LEP-ETU metabolism, including CYP3A4 inducers and inhibitors within 3 weeks prior to, or while receiving, study drug (Please refer to http://medicine.iupui.edu/flockhart/ for a list of such agents).
* Requiring immediate palliative treatment of any kind including surgery and/or radiotherapy.
* Female patients who are pregnant or breast feeding.
* Unwilling or unable to follow protocol requirements.
* Any condition which, in the Investigator's opinion, deems the patient an unsuitable candidate to receive study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48
Dates: Start 2004-11; Primary Completion 2006-11 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
To determine whether LEP-ETU and Taxol are bioequivalent.

SECONDARY OUTCOMES:
To evaluate the pharmacokinetics of paclitaxel and major metabolites in plasma
To assess the safety and tolerability of paclitaxel following intravenous administration of LEP-ETU and Taxol.

CONTACTS AND LOCATIONS:
Locations (6):
- Cancer Institute of New Jersey - University of Medicine and Dentistry of New Jersey, New Brunswick, New Jersey, United States
- Germany (2):
  - Universitatsklinikum Essen, Essen
  - Allgemeines Krankenhaus St. Georg, Hamburg
- Netherlands (3):
  - Academisch Medisch Centrum, Amsterdam
  - Catharina ziekenhuis, Eindhoven
  - Leids Universitair Medisch Centrum, Leiden